CLINICAL TRIAL: NCT05451992
Title: Beneficial Effect of Mediterranean (MD) Components on the Structure and Functions of Gut Microbiome and Metabolome in Subjects With Low Adherence to MD
Brief Title: Microbiome-Tailored Food Products Based On Typical Mediterranean Diet Components
Acronym: SUPERFOOD 19-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, MD, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SuperFood 01
Record Dates: First submitted 2022-06-23; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Microbiota; Overweight and Obesity; Metabolic Complication
Keywords: Microbiota; Mediterranean diet; Overweight; Metabolic syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Control group that will consume a placebo product
  Interventions: Dietary Supplement: Placebo
- SuperFood (Experimental): The superfood group will have to consume the superfood product (vegetable smoothie)
  Interventions: Dietary Supplement: SuperFood

INTERVENTIONS:
Dietary Supplement: Placebo — The group will have to consume a jar every day (approx. 75 ml) which contain (water, malt-dextrins, 0.1% starch, 0.1% guar gum, flavorings and colorants)
  Arms: Placebo
Dietary Supplement: SuperFood — The group will have to consume a jar of superfood (vegetable smoothie) every day. The jar will be filled with approx. 75 ml which corresponds to about 75 g. The superfood formulated by the University of Bolzano on the basis of the results and evidence acquired in collaboration with the Istituto Superiore di Sanità. Composition: pomegranate, walnuts, moringa, broccoli, according to the proportions indicated in Annex 2. This mixture has been analyzed by an external laboratory and authorized for human use
  Arms: SuperFood

SUMMARY:
The composition and functions of the microbiome impact human metabolism and health status. Diet plays a fundamental role in shaping the structure of the gut microbiome, modulating the interaction between the gut microbiome and the human host. Western dietary patterns including a high consumption of red and processed meat, refined grains and sugars, and dairy products have been associated with a high incidence of chronic diseases. It is widely recognised that there is a higher consumption of plant-based foods in Mediterranean countries than in other Western countries. The Mediterranean diet involves a high intake of fruits, vegetables, legumes, nuts, minimally processed cereals, moderate consumption of fish and a low consumption of saturated fats, meat and dairy products with regular intake of extra virgin olive oil. The Mediterranean diet reduces the incidence of cardiovascular, metabolic and neurodegenerative diseases. Interesting results emerged from the evaluation of the microbiome-metabolome interaction, which shows that individuals with the highest adherence to the Mediterranean diet had much higher levels of short-chain fatty acids (SCFAs) and increased levels of the beneficial fiber-degrading bacteria compared to subjects with low adherence to the Mediterranean diet. The study of the effect on the microbiota of specific foods with anti-inflammatory/antioxidant properties is interesting and of potential clinical impact.

DETAILED DESCRIPTION:
The composition and functions of the microbiome impact human metabolism and health status. Dietary habits play a fundamental role in shaping the structure of the gut microbiome, modulating the interactions between the gut microbiome and the human host. Western dietary patterns, including a high consumption of red and processed meat, refined grains and sugars, and dairy products, have been associated with a high incidence of chronic diseases. It is widely recognised that there is a higher consumption of plant-based foods in Mediterranean countries than in other Western countries. The Mediterranean diet involves a high intake of fruits, vegetables, legumes, nuts, minimally processed cereals, moderate consumption of fish and a low consumption of saturated fats, meat and dairy products with regular intake of extra virgin olive oil. The Mediterranean diet (MD) reduces the incidence of cardiovascular, metabolic and neurodegenerative diseases. Interesting results emerged from the evaluation of the microbiome-metabolome interaction, which shows that individuals with the highest adherence to the Mediterranean diet had much higher levels of short-chain fatty acids (SCFAs) and increased levels of the beneficial fiber-degrading bacteria compared to subjects with low adherence to the Mediterranean diet. The study of the effect on the microbiota of specific foods with anti-inflammatory/antioxidant properties is interesting and of potential clinical impact.

Extent and evaluation of current knowledge directly linked to the scientific question(s) to be answered by the clinical study: The Mediterranean diet exerts beneficial effects on health status. Evidence has shown that the two mechanisms by which consuming a Mediterranean diet patterns may contribute to improved metabolic health are modulation of the gastrointestinal microbiota and reduction of metabolic endotoxemia.

Outcomes (efficacy, safety) of completed and number of ongoing clinical studies utilising the same intervention in the same indication: The available evidence focuses on a broader concept of food and nutrient consumption, which do not consider that the beneficial effect of the Mediterranean Diet might due to the synergic and interactive combinations of nutrients, rather than to isolated nutrients.

Level of evidence related to the mechanism of action of the intervention in the planned clinical study population: Although several studies have shown the effects of Mediterranean dietary pattern on health status by modulating intestinal microbiota, a comprehensive evaluation of the synergetic and combined effects of selected dietary pattern on metabolic patterns as well as on the intestinal microbiota and its metabolites is still not totally clarified and recognized.

Objective(s) of the clinical study:

* Primary objective: to explore the effect of a "SuperFood" based on Mediterranean diet components (e.g. dietary fibre, polyphenols, flavonoids and glucosinolates) on the structure and functions of the gut microbiome (bacteria, fungi and viruses) and on the metabolome in subjects with low adherence to Mediterranean Diet.
* Secondary objectives: to explore the effect of a "SuperFood" based on Mediterranean diet components (e.g. dietary fibre, polyphenols, flavonoids and glucosinolates) on the metabolic, inflammatory, and oxidative status, and to define taxonomic and metabolic differences.

Characteristics of the study population (size, age group, sex distribution, inclusion and exclusion criteria; all items with justification!):

Upon signing of the informed consent, 40 healthy volunteers (20 subjects in placebo group and 20 subjects in SuperFood treatment group, comparable sex ratio) with BMI<30 kg/m2 and with low adherence to Mediterranean diet will be enrolled.

Inclusion Criteria:

* Subjects able to sign the Informed Consent
* Age 30-60 years;
* BMI 25-29.9 kg/m2
* Low adherence to the Mediterranean diet (adherence score between 0-5)

Exclusion Criteria:

* Subjects not able to provide informed consent
* obesity (BMI> 30 kg /m2), diabetes, altered thyroid function, food allergies, intestinal disease, liver, kidney, or other organ/apparatus pathologies, regular use of drugs or food supplements, consumption of antibiotics in the 3 months prior to the experiment or need for a specific diet, pregnancy /lactation.
* SARS-CoV-2 infection

Details on sample size and power calculation:

The investigatres considered that a sample of 120 healthy subjects gives sufficient power to detect significant differences regarding certain bacterial strains and metabolites following the consumption of Mediterranean diet components, considering that during the intervention there could be a drop-out rate of 20%.

Design of the clinical study (controlled / uncontrolled; randomised; open / blinded; parallel group / cross over / other; please justify the appropriateness of the selected design) A blinded- and placebo-controlled randomized clinical study of 8 weeks evaluating the possible beneficial effects of a well-selected Mediterranean diet components. Subjects will be randomly assigned to a SuperFood or placebo (blinded) treatment in a 1:1 ratio.

Type of intervention:

The intervention consists of consumption of SuperFood" based on Mediterranean diet components (e.g., dietary fibre, polyphenols, flavonoids and glucosinolates).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to sign the Informed Consent
* Age 30-60 years;
* BMI 25-29.9 kg/m2
* Low adherence to the Mediterranean diet (score between 0-5)

Exclusion Criteria:

* Subjects not able to provide informed consent
* obesity (BMI> 30 kg /m2), diabetes, dysthyroidism, food allergies, alterations of the alvo, any intestinal disease, liver, kidney, or other organ/apparatus pathologies, regular use of drugs or food supplements, consumption of antibiotics in the 3 months prior to the experiment or need for a specific diet, pregnancy /lactation.
* SARS-CoV-2 infection

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Effects of SuperFood on gut Microbiota and metabolome | 2 months
  Analysis of the gut microbiome by DNA extraction from faecal samples and high-throughput rRNA gene-targeted amplicon sequencing Gut metabolome: Faecal samples will be analysed by GC-MS and 1H-NMR. Faecal phenolic compounds and their derivatives as well as endocannabinoids will be also analysed. The amount of faecal SCFA before/after dietary intervention will be used as markers for selecting individuals for further meta-proteomic analysis

SECONDARY OUTCOMES:
Effects of SuperFood on Body Mass Index | 2 months
  height and weight will be combined to calculate Body Mass Index (BMI, expressed as Kg/m^2). measurements will be recorded in all subjects at enrollment and at the end of follow-up
Effects od SuperFood on serum gluco-lipid profile | 2 months
  Serum glucose (mg/dL), total cholesterol (mg/dL), LDL cholesterol (mg/dL), HDL cholesterol (mg/dL), triglycerides (mg/dL) will be measured at enrollment and at the end of the follow-up
Effects of SuperFood on hormones | 2 months
  Serum levels of adiponectin, leptin, insulin, and glucagone will be measured at enrollment and at the end of the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vacca M, Celano G, Calabrese FM, Portincasa P, Gobbetti M, De Angelis M. The Controversial Role of Human Gut Lachnospiraceae. Microorganisms. 2020 Apr 15;8(4):573. doi: 10.3390/microorganisms8040573. PMID 32326636
- [Background] De Angelis M, Garruti G, Minervini F, Bonfrate L, Portincasa P, Gobbetti M. The Food-gut Human Axis: The Effects of Diet on Gut Microbiota and Metabolome. Curr Med Chem. 2019;26(19):3567-3583. doi: 10.2174/0929867324666170428103848. PMID 28462705
- [Background] Vitellio P, Celano G, Bonfrate L, Gobbetti M, Portincasa P, De Angelis M. Effects of Bifidobacterium longum and Lactobacillus rhamnosus on Gut Microbiota in Patients with Lactose Intolerance and Persisting Functional Gastrointestinal Symptoms: A Randomised, Double-Blind, Cross-Over Study. Nutrients. 2019 Apr 19;11(4):886. doi: 10.3390/nu11040886. PMID 31010241
- [Background] Bonfrate L, Di Palo DM, Celano G, Albert A, Vitellio P, De Angelis M, Gobbetti M, Portincasa P. Effects of Bifidobacterium longum BB536 and Lactobacillus rhamnosus HN001 in IBS patients. Eur J Clin Invest. 2020 Mar;50(3):e13201. doi: 10.1111/eci.13201. Epub 2020 Feb 12. PMID 31960952
- [Background] Portincasa P, De Angelis M, Lammert F, Stokes CS. Medicinal Diets: From Molecules to Nutrients to Foods: Basic and Clinical Implications. Curr Med Chem. 2019;26(19):3372-3375. doi: 10.2174/092986732619190821150547. PMID 31564245
- [Background] Portincasa P, Bonfrate L, Vacca M, De Angelis M, Farella I, Lanza E, Khalil M, Wang DQ, Sperandio M, Di Ciaula A. Gut Microbiota and Short Chain Fatty Acids: Implications in Glucose Homeostasis. Int J Mol Sci. 2022 Jan 20;23(3):1105. doi: 10.3390/ijms23031105. PMID 35163038